CLINICAL TRIAL: NCT05684835
Title: Radiographic Prediction of the Nerve Origin of Neck Peripheral Nerve Sheath Tumors: Retrospective Cohort Study
Brief Title: Radiographic Prediction of the Nerve Origin of Neck Peripheral Nerve Sheath Tumors
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Principal Investigator, Chi Chen Huang, Attending doctor, National Cheng-Kung University Hospital
Other Study IDs: A-ER-109-209
Record Dates: First submitted 2023-01-05; First posted 2023-01-13 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Peripheral Nerve Sheath Tumors; Schwannoma of Neck
MeSH Terms: conditions — Nerve Sheath Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Vagus nerve tumor group: patients with neck peripheral nerve sheath tumors originating from the vagus nerve
  Interventions: Procedure: Excision
- Sympathetic nerve tumor group: patients with neck peripheral nerve sheath tumors originating from the sympathetic nerve
  Interventions: Procedure: Excision
- Cervical spinal nerve tumor group: patients with neck peripheral nerve sheath tumors originating from the cervical spinal nerve
  Interventions: Procedure: Excision

INTERVENTIONS:
Procedure: Excision — All patients underwent surgery under general anesthesia and intraoperative neuromonitoring according to the preoperatively predicted NO. Using an anterior cervical approach, the tumor was delineated after identifying the relationships among the great vessels, nerves, and tumors. The NO was confirmed intraoperatively. Sharp dissection was performed meticulously to enucleate the tumor from the NO to preserve most nerve fibers.

SUMMARY:
Postoperative nerve palsy is a major complication following resection of neck peripheral nerve sheath tumors. This study is a retrospective cohort aimed to predict the nerve origin of neck peripheral nerve sheath tumors. Accurate preoperative identification of the nerve origin can improve surgical outcomes and patient counseling

DETAILED DESCRIPTION:
Postoperative nerve palsy is a major complication following resection of neck peripheral nerve sheath tumors (PNSTs). Accurate preoperative identification of the nerve origin (NO) can improve surgical outcomes and patient counseling. This study aims to predict the NO of neck PNSTs with radiographic analysis. This study is a retrospective cohort analysis. Radiographic parameters will be reviewed and the sensitivity, specificity, accuracy of NO prediction will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinical diagnosis of neck peripheral nerve sheath tumors.
* Patients received surgery January 2008 and December 2022.
* The nerve origin of peripheral nerve sheath tumor must be intraoperatively confirmed.

Exclusion Criteria:

* Previous anterior neck surgery.
* Malignant disease.
* Prior neck radiation.
* Undetermined intraoperative nerve origin.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with an intraoperatively confirmed neck PNST and NO between January 2008 and December 2022 who underwent surgical excision of neck PNST with anterior approach, excluding patients with previous anterior neck surgery, malignant disease, prior neck radiation, and undetermined intraoperative NO.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2008-01-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Nerve origin | within 1 month
  intraoperative identification of the nerve origin of the tumor

CONTACTS AND LOCATIONS:
Locations (1):
- National Cheng-Kung University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wong CE, Huang CC, Chuang MT, Lee PH, Chen LY, Hsu HH, Huang CY, Wang LC, Lee JS. Quantification of vessel separation using the carotid-jugular angle to predict the nerve origin of neck peripheral nerve sheath tumours: a pooled analysis of cases from the literature and a single-center cohort. Int J Surg. 2023 Sep 1;109(9):2704-2713. doi: 10.1097/JS9.0000000000000491. PMID 37204443